CLINICAL TRIAL: NCT03042260
Title: Prophylactic Trimethoprim-Sulfamethoxazole for the Prevention of Serious Infections in Patients With Systemic Lupus Erythematosus: a Randomized Placebo Controlled Trial
Brief Title: Prophylactic Trimethoprim/Sulfamethoxazole to Prevent Severe Infections in Patients With Lupus Erythematous
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Jennifer M. Cuellar-Rodríguez, Medical Sciences Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INF-2056-17/20-1
Record Dates: First submitted 2017-01-10; First posted 2017-02-03 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2018-08

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: trimethoprim, sulfamethoxazole drug combination; Infection; Prophylaxis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trimethoprim-Sulfamethoxazole (TMP-SMX) (Experimental): Trimethoprim-Sulfamethoxazole 180mg/800mg oral tablet, 3 times a week, for 6 months. Subjects may remain on the drug longer (maximum 1 year), if they continue to receive intermediate or high dose steroids at the end of 6 months.
  Interventions: Drug: Trimethoprim-Sulfamethoxazole
- Placebo (Placebo Comparator): Tablets that look exactly the same as the experimental drug, 3 times a week, for 6 months.
  Subjects may remain on the placebo longer (maximum 1 year), if they continue to receive intermediate or high dose steroids at the end of 6 months.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Trimethoprim-Sulfamethoxazole — oral tablets, 3 times a week, for a minimum of 6 months and maximum of 1 year.
  Arms: Trimethoprim-Sulfamethoxazole (TMP-SMX)
Drug: Placebo Oral Tablet — oral tablets, 3 times a week, for a minimum of 6 months and maximum of 1 year.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether trimethoprim/sulfamethoxazole is effective in preventing serious infectious complications (those that require hospitalization or lead to death) in patients with lupus erythematosus that receive intermediate or high dose steroids.

ELIGIBILITY:
Inclusion Criteria:

* Systemic Lupus Erythematosus according to the American College of Rheumatology Criteria
* On a daily dose of prednisone of ≥ 15 mg/d or equivalent, and that are expected to remain on the this dose for at least 1 month.
* Have signed an informed consent

Exclusion Criteria:

* Absolute contraindication to receive TMP-SMX (known allergy to TMP-SMX or sulfa drugs; TMP-SMX induced thrombocytopenia)
* Received TMP-SMX treatment in the previous month
* Creatinine clearance <30ml/min/m2
* Chronic viral infection (Hepatitis C virus, Hepatitis B virus, Human immunodeficiency virus)
* Malignant neoplasm, except for skin neoplasm
* Primary immune deficiencies
* Solid organ or hematopoietic stem cell transplant recipients
* Pregnancy or Breastfeeding
* Current active infection, except mild active infections that to the judgement of the primary investigator do not jeopardize the study outcomes (e.g. tinea).
* Uncontrolled chronic infection (e.g. tuberculosis- intensive phase treatment), except mild active chronic infections that to the judgement of the primary investigator do not jeopardize the study outcomes (e.g. onychomycosis).
* Controlled chronic infection, that needs to be treated or prevented with TMP-SMX.
* Absolute Neutrophil Count < 750/mm3, platelets <30x10^9/L, o hemoglobin <7 g/dL
* Patients receiving Methotrexate
* Patients participating in another research study that to the judgement of the principal investigator could jeopardize the safety or efficacy of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of non-viral severe infections | Time on the intervention (maximum 1 year)
  Infections that lead to hospitalization for >24 hours or lead to death.

SECONDARY OUTCOMES:
Serious Adverse Events | Time on the intervention (maximum 1 year)
  A serious adverse event is an adverse event that leads to death, persistent disability, leads to hospitalization or increase in length of hospitalization. Additionally, an adverse event that does not immediately put life at risk, but that requires a medical or surgical intervention to prevent a serious adverse event.
Frequency of non-viral infections | Time on the intervention (maximum 1 year)
  All non-viral infections (severe and non-severe)
Time to first episode of non-viral severe infection | From 2 weeks after randomization until the date of the first episode of a non-viral severe infection, up to 1 year after randomization.
  Infections that lead to hospitalization for >24 hours or lead to death, that are not of viral etiology.
All cause mortality or hospitalization | Time on the intervention (maximum 1 year)
  Death or hospitalization due to any cause infectious or non-infectious
Proportion of patients that develop infections resistant to TMP-SMX | Time on the intervention (maximum 1 year)
  Infections that would traditionally be considered susceptible to TMP-SMX
Drug discontinuation | 1 year
  Number of patients that require drug discontinuation due to safety concerns

OTHER OUTCOMES:
Peripheral Blood Immunophenotype: B and T lymphocytes and Natural Killer (NK) cells measured by multiparametric flow cytometry. These variables will be expressed as % of total peripheral blood mononuclear cells (PBMC) | Up to 1 year after randomization.
  In a random sample of a subset of patients, serially examined parameters at baseline, development of a first episode of severe infection or at the end of follow-up. Variables will be described as mean and standard deviation and groups will be compared by means of student T test. Association will be assessed by ANCOVA.
Peripheral Blood Immunophenotype: Absolute number of B and T lymphocytes and NK cells per mcl of blood, measured by multiparametric flow cytometry. | Up to 1 year after randomization.
  In a random sample of a subset of patients, serially examined parameters at baseline, development of a first episode of severe infection or at the end of follow-up. Variables will be described as mean and standard deviation and groups will be compared by means of student T test. Association will be assessed by ANCOVA.
Innate Immune Cells Phagocytosis: Mean fluorescence intensity of (pHrodo) positive cells. | Up to 1 year after randomization
  In a random sample of a subset of patients, serially examined parameters at baseline, development of a first episode of severe infection or at the end of follow-up. Variables will be described as mean and standard deviation and groups will be compared by means of student T test. Association will be assessed by ANCOVA.
Innate Immune Cells Phagocytosis:Percentage of (pHrodo) positive cells. | Up to 1 year after randomization
  In a random sample of a subset of patients, serially examined parameters at baseline, development of a first episode of severe infection or at the end of follow-up. Variables will be described as mean and standard deviation and groups will be compared by means of student T test. Association will be assessed by ANCOVA.
Respiratory Burst from Neutrophils by dihydrorhodamine; expressed as mean fluorescence intensity. | Up to 1 year after randomization
  In a random sample of a subset of patients, serially examined parameters at baseline, development of a first episode of severe infection or at the end of follow-up. Variables will be described as mean and standard deviation and groups will be compared by means of student T test. Association will be assessed by ANCOVA.
Respiratory Burst from Neutrophils by dihydrorhodamine; expressed as percentage of positive cells. | Up to 1 year after randomization
  In a random sample of a subset of patients, serially examined parameters at baseline, development of a first episode of severe infection or at the end of follow-up. Variables will be described as mean and standard deviation and groups will be compared by means of student T test. Association will be assessed by ANCOVA.
Neutrophil Extracellular Traps (NETs): Mean fluorescence of Sytox Green by spectrometry from lipopolysaccharide stimulated neutrophils. | Up to 1 year after randomization
  In a random sample of a subset of patients, serially examined parameters at baseline, development of a first episode of severe infection or at the end of follow-up. Variables will be described as mean and standard deviation and groups will be compared by means of student T test. Association will be assessed by ANCOVA.
Neutrophil Extracellular Traps (NETs): Normalized mean fluorescence of elastase and Hoechst in 6 optical fields for each sample. | Up to 1 year after randomization
  In a random sample of a subset of patients, serially examined parameters at baseline, development of a first episode of severe infection or at the end of follow-up. Variables will be described as mean and standard deviation and groups will be compared by means of student T test. Association will be assessed by ANCOVA.
Changes in systemic lupus erythematosus (SLE) activity using SLEDAI (Lupus Erythematosus Activity Index ) | Up to 1 year after randomization
  Serially calculated over time at standard 3 months intervals (determined as mild, moderate or severe activity)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Cuellar-Rodriguez, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Background] Danza A, Ruiz-Irastorza G. Infection risk in systemic lupus erythematosus patients: susceptibility factors and preventive strategies. Lupus. 2013 Oct;22(12):1286-94. doi: 10.1177/0961203313493032. PMID 24098001
- [Background] Cervera R, Khamashta MA, Font J, Sebastiani GD, Gil A, Lavilla P, Mejia JC, Aydintug AO, Chwalinska-Sadowska H, de Ramon E, Fernandez-Nebro A, Galeazzi M, Valen M, Mathieu A, Houssiau F, Caro N, Alba P, Ramos-Casals M, Ingelmo M, Hughes GR; European Working Party on Systemic Lupus Erythematosus. Morbidity and mortality in systemic lupus erythematosus during a 10-year period: a comparison of early and late manifestations in a cohort of 1,000 patients. Medicine (Baltimore). 2003 Sep;82(5):299-308. doi: 10.1097/01.md.0000091181.93122.55. PMID 14530779
- [Background] Barber C, Gold WL, Fortin PR. Infections in the lupus patient: perspectives on prevention. Curr Opin Rheumatol. 2011 Jul;23(4):358-65. doi: 10.1097/BOR.0b013e3283476cd8. PMID 21532484
- [Background] Bwakura-Dangarembizi M, Kendall L, Bakeera-Kitaka S, Nahirya-Ntege P, Keishanyu R, Nathoo K, Spyer MJ, Kekitiinwa A, Lutaakome J, Mhute T, Kasirye P, Munderi P, Musiime V, Gibb DM, Walker AS, Prendergast AJ. A randomized trial of prolonged co-trimoxazole in HIV-infected children in Africa. N Engl J Med. 2014 Jan 2;370(1):41-53. doi: 10.1056/NEJMoa1214901. PMID 24382064
- [Background] Vananuvat P, Suwannalai P, Sungkanuparph S, Limsuwan T, Ngamjanyaporn P, Janwityanujit S. Primary prophylaxis for Pneumocystis jirovecii pneumonia in patients with connective tissue diseases. Semin Arthritis Rheum. 2011 Dec;41(3):497-502. doi: 10.1016/j.semarthrit.2011.05.004. Epub 2011 Sep 29. PMID 21959291